CLINICAL TRIAL: NCT06110234
Title: Interindividual Variability in Cognitive Aging: Neural Mechanisms, Reserve Processes and Malleability of Neuroprotective Processes.
Brief Title: Efficacy, Transfer, and Neuro-functional Basis of a Memory Training Targeting Episodic Retrieval in Older Adults.
Acronym: SPECTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Sylvie Belleville, Principal Investigator, Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CRIUGM-007
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: Memory, Episodic; Aging; Cognitive Training; Transfer, Psychology; Neuropsychology; Cognitive Psychology; Neurosciences
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Intervention Model Description: Older participants are randomly assigned to one of two intervention conditions (Episodic Specificity Induction ; Associative Memory)
Who Masked: Participant, Outcomes Assessor
Masking Description: Assessors are blind in the clinical trials. Participants know that there are different training programs but they ignore the purpose of each one.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Episodic Specificity Induction (Experimental): In each of the six training sessions, participants practice the ESI first under supervision and then unsupervised (self-administered). Self-administration is performed on a laptop. During each practice of the ESI, participants perform a detailed recall of a new 1-minute video clip of a complex scene - a skit of the famous English comedian Mr. Bean. Each session lasts for 90 minutes.
  Interventions: Behavioral: Episodic Specificity Induction
- Associative Memory (Active Comparator): In each of the six training sessions, participants recall pairs of words and pictures (e.g., names of women and rings). These pairs are presented successively after a fictitious scenario is presented to motivate memorization. There are 12 scenarios, each with 5 different word/picture pairs. Simple additions and subtractions separate the encoding phase from the recall phase. This training is adapted from Bellander et al, (2017). A general knowledge quiz is also administered at the end of the session. The training is performed on a laptop. Each session lasts for 90 minutes.
  Interventions: Behavioral: Associative Memory

INTERVENTIONS:
Behavioral: Episodic Specificity Induction — Recalling complex scenes using the Episodic Specificity Induction
  Arms: Episodic Specificity Induction
Behavioral: Associative Memory — Recalling word/picture pairs
  Arms: Associative Memory

SUMMARY:
Aging leads to cognitive changes that affect memory, particularly episodic retrieval. These impairments are detrimental to seniors' quality of life. Cognitive trainings are of great interest to the scientific community because they improve cognition in older people, and produce structural and functional changes likely to provide neuroprotection. Identifying the brain changes induced by cognitive training could therefore provide a better understanding of the neuroplastic processes of the aging brain. Some training programs aim to improve key processes underlying cognitive functioning to lead to transfer, but these most often target working memory or processing speed. Our aim is to understand the brain changes associated with a training program targeting episodic retrieval, and likely to engage a core network for memory, including the anterior hippocampus. 60 healthy older adults will be randomly divided into two groups; one receiving a training based on the Episodic Specificity Induction (ESI) - a manipulation based on a well-established police interviewing technique thought to target and facilitate episodic construction; the other receiving a control training consisting of recalling pairs of words and images. Before and after training, behavioural and brain measures will be taken. Behavioural measures will be taken during recall, recognition, and problem solving tasks. These tasks will be completed once in the ESI condition (after one ESI) and once in the NoESI condition (after a general thoughts interview). Measures of brain activation as well as static and dynamic functional connectivity (SFC & DFC) will be taken using magnetic resonance imaging (MRI) during a recognition task. For behavioural measures, higher pre-training performance should be observed in the ESI than in the NoESI condition, and pre-to-post-training improvement should be observed only after the ESI training, especially in the NoESI condition. For brain measures, ESI training should decrease activation of the task network targeted by training, reflecting an increase in efficiency. ESI training should also increase the SFC of the task network and reduce its connectivity with the cognitive control network, suggesting more automated processing. Finally, ESI training should increase DFC by increasing the speed of transition between the networks associated with the two phases of episodic retrieval: the construction phase and the elaboration phase.

DETAILED DESCRIPTION:
Aging leads to cognitive changes that affect memory, particularly episodic retrieval, which is involved in remembering an event within a specific spatio-temporal context. These impairments are detrimental to seniors' quality of life. Recently, cognitive training has attracted considerable interest in the scientific community, as it improves cognition in older adults, and produces structural and functional changes. They are considered a form of "late education" likely to provide neuroprotection. A better understanding of training-induced brain changes is therefore essential to a better understanding of the neuroplastic potential of the aging brain. A distinction is made between training that aims to teach strategies, and training that aims to repeatedly practice a task that involves a key process to facilitate it. The latter are recognized as having greater potential to induce a transfer of their benefits to untrained abilities. According to the INTERACTIVE model, they would lead to a decrease in activation in the brain regions involved in the task, due to more efficient processing within specialized regions. Yet there are very few training programs that target episodic retrieval. Developing such trainings would therefore contribute to our understanding of training-induced brain changes. One key process involved in episodic retrieval that such training could target is scene construction. This corresponds to the ability to mentally generate and maintain the coherence of a complex scene. It would engage the anterior hippocampus, especially its medial part, and a "core" network comprising the medial temporal lobes, parahippocampal cortex, and posterior parietal regions such as the retrosplenial cortex and precuneus. Studies suggest that this process may be targeted and facilitated when participants are interviewed about their memory of a video via an Episodic Specificity Induction (ESI) - a manipulation based on a well-established police interviewing technique knwon as the Cognitive Interview (CI). This technique promotes mental imagery, structures recall, and emphasizes spatial relationships between entities in a scene. At the behavioral level, it has been shown in both young and old adults that receiving a single ESI just before performing a task of interest involving scene construction temporarily improves performance on that task. At the brain level, the ESI has been shown in young adults to increase activation of brain regions involved in scene construction during the task of interest, specifically during the construction phase. This phase corresponds to the retrieval of the event representation, and precedes the elaboration phase, associated with the retrieval of additional details (see construction-elaboration paradigm). These two phases have common and distinct neural correlates. The construction phase is associated with stronger connectivity of the left anterior hippocampus with the right anterior hippocampus and left frontotemporal regions, while the elaboration phase is associated with stronger connectivity of the left anterior hippocampus with the bilateral posterior hippocampus and visual perception regions. However, the ESI has never been adapted within a training program to study its effects on the aged brain. In a proof-of-concept study, we tested on 16 healthy older adults an ESI-based training program that we co-created with potential future end-users. We observed transfer to free recall and recognition tasks, but also to a problem-solving and divergent creative thinking tasks, which are not purely memory tasks, but which would involve scene construction. In the present study, we aim to compare the ESI-based training with an active control training and investigate the neural substrates involved.

60 healthy older adults (60-85 years) will be recruited for this study. All participants will be recruited from the community and living in the Montreal area. A telephone interview will provide initial selection information. Eligible persons will be invited to come to the laboratory for a short neuropsychological assessment to evaluate their clinical status and cognitive functioning, as well as a behavioural assessment (PRE). Concerning behavioural tasks, three tasks from the proof-of-concept study will be used: free recall and recognition (as nearest- and near-transfer outcomes) and problem solving (as far-transfer outcome). These tasks will be completed twice, once in the ESI condition right after receiving one ESI; once in the NoESI condition right after receiving a general thoughts interview. Behavioural assessment session will last 2 hours. The pre-training behavioural assessment session will be followed on average two days later by a functional magnetic resonance imaging (fMRI) scan. Concerning the fMRI task: outside the scan, participants will first encode short videos of scenes from everyday life along with their titles. Then, in the scan, each title will be presented and participants will answer questions about the spatial relationships between objects that were present in the video associated with the title. The fMRI sessions will last 1 hour (including 30 minutes in the scanner). Participants will be randomly assigned to one of two training groups (ESI vs. Active control). The ESI-based training consists in recalling short video clips using the ESI, first supervised, then unsupervised (self-administered). The active control training consists in recalling associations between pictures and words. Participants will be trained in small groups of 4 individuals, for a total of 15 groups. On average, outcome measures will be taken a week prior the first training session (PRE), and the day after the last training session (POST). Different version of the tasks will be used in the pre- and post training assessment, as well as, in the ESI and NoESI conditions.

The effect of training on behavioural measures will be assessed. For the three tasks (free recall, recognition and problem solving), higher pre-training performance should be observed in the ESI than in the NoESI condition, and pre-to-post-training improvement should be observed only after the ESI training, especially in the NoESI condition. The effect of training on brain activation and static and dynamic functional connectivity (SFC & DFC) will also be assessed. Concerning brain activation, activation of the medial temporal lobe during the construction phase, and especially the left anterior hippocampus and inferior parietal lobe involved in scene construction, should decrease after the ESI training, suggesting an increase in brain efficiency. For static FC, the ESI training should increase the modularity of the core brain network related to episodic processing, including the hippocampus, bilateral parahippocampal gyrus, angular gyrus, medial prefrontal cortex, precuneus and retrosplenial/posterior cortex. It should also reduce communication with the fronto-parietal brain network related to cognitive control (i.e., bilateral lateral prefrontal cortex, anterior cingulate and precuneus), reflecting greater segregation and more automated processing. For dynamic FC, we will look at temporal reconfigurations of FC within and between task-associated networks, before and after training. ESI-trained participants should be faster to switch from an integrated network for the construction phase, to an integrated network for the elaboration phase, suggesting an adaptation of cognitive processing strategies.

ELIGIBILITY:
Inclusion Criteria:

* French-speaking
* Right-handed
* Sufficient visual and auditory acuity to undergo neuropsychological tests and to do the interventions.
* Sufficient delayed recall score above the education-adjusted cut-offs (≥9 for 16+ years of education; ≥5 for 8-15 years of education; ≥3 for 0-7 years of education) at the Logical Memory test (Wechsler Memory Scale, maximum score 25).

Exclusion Criteria:

* A score bellow the education-adjusted cut-offs at the MoCA ( <24 for >12 years of education; <23 for = or <12 years of education)
* Answer 'Yes' to the two following questions: "Do you feel like your memory is becoming worse?" "Does this worry you?" (to exclude subjective cognitive decline).
* The presence of a disease or injury of the central nervous system: moderate to severe chronic static leukoencephalopathy (including previous traumatic injury), multiple sclerosis, a serious developmental handicap, subdural hematoma (past or current), subarachnoid haemorrhage (past or current), primary cerebral tumour or cerebral metastases, epilepsy (current), dementia or another neurodegenerative disease, and other rarer brain illnesses.
* Symptomatic stroke within the previous year.
* Alcoholism or substance abuse
* History of intracranial surgery.
* Major surgery within last 2 months.
* General anesthesia in the past 6 months.
* Serious comorbid condition that, in the opinion of the study investigator, is likely to result in death within a year.
* Major depression or anxiety.
* Schizophrenia or other major psychiatric disorder (e.g., bipolar disorder).
* Individuals where French is not sufficiently proficient for clinical assessment and neuropsychological testing.
* Unable to undergo MRI scan due to medical contraindications or inability to tolerate the procedure.
* Plans on moving outside the province within the next 2 months.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Changes in the number of correct specific detail recall (nearest transfer outcome) | In the week preceding the start of the intervention (PRE) both in the ESI and the NoESI condition; In the week of the last intervention session (POST) both in the ESI and the NoESI condition
  For the free recall task, verbal recall will be recorded and transcribed. Recalled details will be rated as specific according to the Autobiographical Interview procedure developed by Levine et al (2002). The number of specific details recalled will be measured, and the accuracy of these details will be evaluated. The number of correct specific details will be calculated by subtracting the incorrect specific details from the recalled specific details. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Brain function: Memory related activation | In the week preceding the start of the intervention (PRE); In the week of the last intervention session (POST)
  Functional activations. Functional images are acquired on a 3.0T Siemens Prisma scanner using 32-channel head coil and Simultaneous multi-slice (SMS) echo planar imaging (EPI) sequence: parallel imaging parameters: multiband factor = 3 with GRAPPA (R) factors 2; TR = 0.910 s; TE = 20 ms; flip angle 56°; voxels 2.5 mm³; 57 slices; FOV: 200; acquisition matrix: 80 x80
Brain function: Memory related activation (Static functional connectivity) | In the week preceding the start of the intervention (PRE); In the week of the last intervention session (POST)
  Static functional connectivity. Functional images are acquired on a 3.0T Siemens Prisma scanner using 32-channel head coil and Simultaneous multi-slice (SMS) echo planar imaging (EPI) sequence: parallel imaging parameters: multiband factor = 3 with GRAPPA (R) factors 2; TR = 0.910 s; TE = 20 ms; flip angle 56°; voxels 2.5 mm³; 57 slices; FOV: 200; acquisition matrix: 80 x80
Brain function: Memory related activation (Dynamic functional connectivity) | In the week preceding the start of the intervention (PRE); In the week of the last intervention session (POST)
  Dynamic functional connectivity. Functional images are acquired on a 3.0T Siemens Prisma scanner using 32-channel head coil and Simultaneous multi-slice (SMS) echo planar imaging (EPI) sequence: parallel imaging parameters: multiband factor = 3 with GRAPPA (R) factors 2; TR = 0.910 s; TE = 20 ms; flip angle 56°; voxels 2.5 mm³; 57 slices; FOV: 200; acquisition matrix: 80 x80
Changes in the measure of discriminability (d') (near transfer outcome) - fMRI | In the week preceding the start of the intervention (PRE); In the week of the last intervention session (POST)
  For the fMRI recognition task, a d' measure will be calculated using the following formula: d' = z(hit rate) - z(false alarm rate). Higher scores mean a better outcome.
Changes in the number of relevant steps produced (far transfer outcome) | In the week preceding the start of the intervention (PRE) both in the ESI and the NoESI condition; In the week of the last intervention session (POST) both in the ESI and the NoESI condition
  For the problem solving task, verbal production of steps will be recorded and transcribed, and the number of relevant steps will be computed using the same procedure as Madore & Schacter (2014). Higher scores mean a better outcome.
Changes in the measure of discriminability (d') (near transfer outcome) | In the week preceding the start of the intervention (PRE) both in the ESI and the NoESI condition; In the week of the last intervention session (POST) both in the ESI and the NoESI condition
  For the recognition task, a d' measure will be calculated using the following formula: d' = z(hit rate) - z(false alarm rate). Higher scores mean a better outcome.

OTHER OUTCOMES:
Effect of moderators: Sex. | In the week preceding the start of the intervention (PRE)
  Male vs Female on the intervention effect
Effect of moderators: Cognitive reserve proxies. | In the week preceding the start of the intervention (PRE)
  Scores on the reserve-proxy questionnaire (from Rami L, Valls-Pedret C, Bartres-Faz D, et al. 2011) on the intervention effect

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Belleville, PhD, Principal Investigator — Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Locations (1):
- CRIUGM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: No more than one year after the end of the data collection.
Access Criteria: Public.
URL: https://osf.io/cwtfp/